CLINICAL TRIAL: NCT02112916
Title: A Phase III Randomized Trial Investigating Bortezomib (NSC# 681239) on a Modified Augmented BFM (ABFM) Backbone in Newly Diagnosed T-Lymphoblastic Leukemia (T-ALL) and T-Lymphoblastic Lymphoma (T-LLy)
Brief Title: Combination Chemotherapy With or Without Bortezomib in Treating Younger Patients With Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia or Stage II-IV T-Cell Lymphoblastic Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00712; NCI-2014-00712 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s14-01925; AALL1231 (Other: Children's Oncology Group); AALL1231 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Adult T Acute Lymphoblastic Leukemia; Ann Arbor Stage II Adult Lymphoblastic Lymphoma; Ann Arbor Stage II Childhood Lymphoblastic Lymphoma; Ann Arbor Stage III Adult Lymphoblastic Lymphoma; Ann Arbor Stage III Childhood Lymphoblastic Lymphoma; Ann Arbor Stage IV Adult Lymphoblastic Lymphoma; Ann Arbor Stage IV Childhood Lymphoblastic Lymphoma; Childhood T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Etoposide; Hydrocortisone; hydrocortisone hemisuccinate; Ifosfamide; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Radiotherapy; Radiation; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (combination chemotherapy) (Active Comparator): Patients receive combination chemotherapy without bortezomib. See Detailed Description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Hydrocortisone Sodium Succinate; Drug: Ifosfamide; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine; Drug: Vincristine Sulfate
- Arm B (combination chemotherapy, bortezomib) (Experimental): Patients receive combination chemotherapy with bortezomib (4 doses at 1.3 mg/m^2 during Induction and 4 doses at 1.3 mg/m^2 during Delayed Intensification). See Detailed Description.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Hydrocortisone Sodium Succinate; Drug: Ifosfamide; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
  Arms: Arm B (combination chemotherapy, bortezomib)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IT, IV, or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Hydrocortisone Sodium Succinate — Given IT
  Other Names: (11beta)-21-(3-Carboxy-1-oxopropyl)-11,17-dihydroxypregn-4-ene-3,20-dione, Monosodium Salt; A-Hydrocort; Buccalsone; Corlan; Cortisol Sodium Succinate; Cortop; Efcortelan; Emergent-EZ; Flebocortid; Hidroc Clora; Hycorace; Hydro-Adreson; Hydrocort; Hydrocortisone 21-Sodium Succinate; Hydrocortisone Na Succinate; Kinogen; Nordicort; Nositrol; Sinsurrene; Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Leucovorin Calcium — Given PO or IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Give PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, IV, or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial compares how well combination chemotherapy works when given with or without bortezomib in treating patients with newly diagnosed T-cell acute lymphoblastic leukemia or stage II-IV T-cell lymphoblastic lymphoma. Bortezomib may help reduce the number of leukemia or lymphoma cells by blocking some of the enzymes needed for cell growth. It may also help chemotherapy work better by making cancer cells more sensitive to the drugs. It is not yet known if giving standard chemotherapy with or without bortezomib is more effective in treating newly diagnosed T-cell acute lymphoblastic leukemia and T-cell lymphoblastic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare event-free survival (EFS) in patients with newly diagnosed T-cell acute lymphoblastic leukemia (T-ALL) and T-cell lymphoblastic lymphoma (T-LLy) who are randomized to a modified augmented Berlin-Frankfurt-Munster (ABFM) backbone versus bortezomib plus the modified ABFM backbone.

SECONDARY OBJECTIVES:

I. To determine the safety and feasibility of modifying standard therapy for T-ALL and T-LLy based on the results of UKALL 2003, which includes a dexamethasone-based induction, additional doses of pegaspargase (PEG-ASP) during induction and delayed intensification (DI), and dexamethasone pulses during maintenance therapy.

II. To determine if prophylactic (presymptomatic) cranial radiation therapy (CRT) can be safely and effectively eliminated in the 85-90% of T-ALL patients classified as standard or intermediate risk.

III. To determine the proportion of end of consolidation (EOC) minimal residual disease (MRD) >= 0.1% T-ALL patients who become MRD negative (undetectable by flow cytometry) after intensification of chemotherapy, using three high risk (HR) BFM blocks, and to compare EFS between the patients who become MRD negative after the three HR BFM blocks and continue on chemotherapy with those who continue to have detectable MRD and are eligible for other treatment strategies, including hematopoietic stem cell transplant (HSCT).

IV. To compare the EFS between very high risk (induction failure) T-LLy patients treated with HR BFM intensification blocks who have partial or complete response (PR or CR) with those who do not respond (NR).

CORRELATIVE OBJECTIVES:

I. To investigate the prognostic significance of day 29 bone marrow (BM) MRD in T-LLy patients.

II. To determine if protein expression patterns can predict bortezomib response and drug resistance in T-ALL.

III. To analyze and target relevant signaling pathways in T-ALL blasts, focusing on early T cell precursor (ETP) acute lymphoblastic leukemia (ALL).

OUTLINE: Patients are randomized to 1 of 2 treatment arms. Patients are risk assigned based on data from end of induction and/or consolidation therapy; this then modifies the subsequent therapy received.

T-ALL Risk Group Definitions:

Standard Risk (SR): CNS1*, lumbar puncture prior to steroid therapy (not steroid pretreated), Day 29 (end of induction) bone marrow M1, Day 29 bone marrow minimal residual disease (MRD) <=0.01%, no testicular leukemia at diagnosis.

Intermediate Risk (IR): Not SR or VHR.

Very High Risk (VHR): M3 marrow at Day 29 and/or end of consolidation (EOC) MRD >=0.1%.

*CNS2 and CNS3 cannot be SR and are assigned to IR or VHR based on marrow response.

T-LL Risk Group Definitions:

Standard Risk (SR): CNS1*, MRD at diagnosis <1% in bone marrow, lumbar puncture prior to steroid therapy (not steroid pretreated), Day 29 (end of induction) complete response (CR) or partial response (PR).

Intermediate Risk (IR): Not SR or VHR.

Very High Risk (VHR): Stable Disease (SD)/No response (NR) at Day 29 (End of Induction).

*CNS2 and CNS3 cannot be SR and are assigned to IR or VHR based on radiographic response.

ARM A INDUCTION: Patients receive cytarabine intrathecally (IT) at time of diagnostic lumbar puncture (if within 72 hours from start of protocol therapy) OR day 1; vincristine sulfate intravenously (IV) over 1 minute on days 1, 8, 15, and 22; dexamethasone orally (PO) twice daily (BID) on days 1-28 (no taper); daunorubicin hydrochloride IV over 1-15 minutes on days 1, 8, 15, and 22; pegaspargase IV over 1-2 hours on days 4 and 18; and methotrexate IT on days 8 and 29 (and on days 15 and 22 for central nervous system 3 involvement [CNS3] T-ALL patients).

ARM A CONSOLIDATION: Beginning on day 36 from Induction, patients receive methotrexate IT on days 1, 8, 15, and 22 (days 1 and 8 only for CNS3 T-ALL or CNS3 T-LLy patients); cyclophosphamide IV over 30-60 minutes on days 1 and 29; cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO once daily (QD) on days 1-14 and 29-42; pegaspargase IV over 1-2 hours on days 15 and 43; and vincristine sulfate IV on days 15, 22, 43, and 50. Patients with persistent testicular disease undergo radiation therapy.

Patients are then assigned to subsequent therapy according to risk assignment. Patients with standard risk (SR) disease receive Interim Maintenance with Capizzi methotrexate (CMTX); patients with intermediate risk (IR) disease receive Interim Maintenance with high-dose methotrexate (HDMTX), Delayed Intensification, and then Interim Maintenance with CMTX; and patients with very high risk (VHR) disease receive 3 HR Intensification Blocks, Delayed Intensification, and then Interim Maintenance with CMTX.

ARM A CMTX INTERIM MAINTENANCE: Patients receive vincristine sulfate IV over 1 minute on days 1, 11, 21, 31, and 41; methotrexate IV over 2-5 minutes (undiluted) or 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41; pegaspargase IV over 1-2 hours on days 2 and 22; and methotrexate IT on days 1 and 31. The next course (based on risk assignment) begins on day 57 or when blood counts recover (whichever occurs later).

ARM A DELAYED INTENSIFICATION: Patients receive vincristine sulfate IV over 1 minute on days 1, 8, 15, 43, and 50; dexamethasone PO BID or IV on days 1-7 and 15-21; doxorubicin hydrochloride IV over 15 minutes on days, 1, 8, and 15; pegaspargase IV over 1-2 hours on days 4, 18, and 43; methotrexate IT on days 1, 29, and 36; cyclophosphamide IV over 30-60 minutes on day 29; cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39; and thioguanine PO on days 29-42. The next course (based on risk assignment) begins on day 64 or when blood counts recover (whichever occurs later).

ARM A HDMTX INTERIM MAINTENANCE: Patients receive high-dose methotrexate IV over 24 hours on days 1, 15, 29, and 43; leucovorin calcium IV or PO on days 3-4, 17-18, 31-32, and 45-46; vincristine sulfate IV on days 1, 15, 29, and 43; mercaptopurine PO QD on days 1-56; and methotrexate IT on days 1 and 29. The next course (based on randomization assignment) begins on day 57 or when blood counts recover (whichever occurs later).

ARM A INTENSIFICATION BLOCK I: Patients receive dexamethasone IV or PO BID on days 1-5; high-dose methotrexate IV over 24 hours on day 1; leucovorin calcium IV or PO on days 3-4; vincristine sulfate IV on days 1 and 6; cyclophosphamide IV over 1-6 hours on days 2-4; high-dose cytarabine IV over 3 hours every 12 hours on day 5; pegaspargase IV over 1-2 hours on day 6; and triple IT therapy comprising methotrexate IT, hydrocortisone IT, and cytarabine IT on day 1. The next course (Intensification Block II) begins on day 22 or when blood counts recover (whichever occurs later).

ARM A INTENSIFICATION BLOCK II: Patients receive dexamethasone PO BID or IV on days 1-5; high-dose methotrexate IV over 24 hours on day 1; leucovorin calcium PO or IV on days 3-4; vincristine sulfate IV on days 1 and 6; ifosfamide IV over 1 hour every 12 hours on days 2-4; daunorubicin hydrochloride IV over 30 minutes on day 5; pegaspargase IV over 1-2 hours on day 6; and triple IT therapy on day 1 as in Intensification Block I. The next course (Intensification Block III) begins on day 22 or when blood counts recover (whichever occurs later).

ARM A INTENSIFICATION BLOCK III: Patients receive dexamethasone PO BID or IV on days 1-5; high-dose cytarabine IV over 3 hours every 12 hours on days 1-2; etoposide IV over 1-2 hours every 12 hours on days 3-5; pegaspargase IV over 1-2 hours on day 6; and triple IT therapy on day 5 as in Intensification Block I. The next course (based on randomization) begins on day 22 or when blood counts recover (whichever occurs later).

ARM A MAINTENANCE THERAPY: All patients receive vincristine sulfate IV over 1 minute on days 1, 29, and 57; dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61; mercaptopurine PO on days 1-84; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (omit day 29 for SR patients during the first 4 cycles); methotrexate IT on day 1 (and day 29 during the first 4 cycles for SR patients and during the first 2 cycles for IR patients). Patients with CNS1-3VHR and CNS2 VHR, and CNS3 IR disease also undergo cranial radiation therapy during the first 4 weeks (cycle 1). Treatment in female patients with T-ALL and patients with T-LLY repeats every 12 weeks for up to 2 years from the start of Interim Maintenance (week 119). Treatment in male patients with T-ALL repeats every 12 weeks for up to 3 years from the start of Interim Maintenance (week 171).

ARM B INDUCTION: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11(1.3 mg/m^2 per dose); and cytarabine, vincristine sulfate, dexamethasone, daunorubicin hydrochloride, pegaspargase, and methotrexate as in Induction Arm A.

ARM B CONSOLIDATION: Beginning on day 36 from Induction, patients receive methotrexate IT on days 1, 8, 15, and 22 (days 1 and 8 only for CNS3 T-ALL or CNS3 T-LLy patients); cyclophosphamide IV over 30-60 minutes on days 1 and 29; cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO once daily (QD) on days 1-14 and 29-42; pegaspargase IV over 1-2 hours on days 15 and 43; and vincristine sulfate IV on days 15, 22, 43, and 50. Patients with persistent testicular disease undergo radiation therapy.

Patients are then assigned to subsequent therapy according to risk assignment. Patients with standard risk (SR) disease receive Interim Maintenance with Capizzi methotrexate (CMTX); patients with intermediate risk (IR) disease receive Interim Maintenance with high-dose methotrexate (HDMTX), Delayed Intensification, and then Interim Maintenance with CMTX; and patients with very high risk (VHR) disease receive 3 HR Intensification Blocks, Delayed Intensification, and then Interim Maintenance with CMTX.

ARM B CMTX INTERIM MAINTENANCE: Patients receive vincristine sulfate IV over 1 minute on days 1, 11, 21, 31, and 41; methotrexate IV over 2-5 minutes (undiluted) or 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41; pegaspargase IV over 1-2 hours on days 2 and 22; and methotrexate IT on days 1 and 31. The next course (based on risk assignment) begins on day 57 or when blood counts recover (whichever occurs later).

ARM B DELAYED INTENSIFICATION: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 15, and 18 (1.3 mg/m^2 per dose); and vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, methotrexate, cyclophosphamide, cytarabine, and thioguanine as in Delayed Intensification Arm A. The next course (based on risk assignment) begins on day 64 or when blood counts recover (whichever occurs later).

ARM B HDMTX INTERIM MAINTENANCE: Patients receive high-dose methotrexate IV over 24 hours on days 1, 15, 29, and 43; leucovorin calcium IV or PO on days 3-4, 17-18, 31-32, and 45-46; vincristine sulfate IV on days 1, 15, 29, and 43; mercaptopurine PO QD on days 1-56; and methotrexate IT on days 1 and 29. The next course (based on randomization assignment) begins on day 57 or when blood counts recover (whichever occurs later).

ARM B INTENSIFICATION BLOCK I: Patients receive dexamethasone IV or PO BID on days 1-5; high-dose methotrexate IV over 24 hours on day 1; leucovorin calcium IV or PO on days 3-4; vincristine sulfate IV on days 1 and 6; cyclophosphamide IV over 1-6 hours on days 2-4; high-dose cytarabine IV over 3 hours every 12 hours on day 5; pegaspargase IV over 1-2 hours on day 6; and triple IT therapy comprising methotrexate IT, hydrocortisone IT, and cytarabine IT on day 1. The next course (Intensification Block II) begins on day 22 or when blood counts recover (whichever occurs later).

ARM B INTENSIFICATION BLOCK II: Patients receive dexamethasone PO BID or IV on days 1-5; high-dose methotrexate IV over 24 hours on day 1; leucovorin calcium PO or IV on days 3-4; vincristine sulfate IV on days 1 and 6; ifosfamide IV over 1 hour every 12 hours on days 2-4; daunorubicin hydrochloride IV over 30 minutes on day 5; pegaspargase IV over 1-2 hours on day 6; and triple IT therapy on day 1 as in Intensification Block I. The next course (Intensification Block III) begins on day 22 or when blood counts recover (whichever occurs later).

ARM B INTENSIFICATION BLOCK III: Patients receive dexamethasone PO BID or IV on days 1-5; high-dose cytarabine IV over 3 hours every 12 hours on days 1-2; etoposide IV over 1-2 hours every 12 hours on days 3-5; pegaspargase IV over 1-2 hours on day 6; and triple IT therapy on day 5 as in Intensification Block I. The next course (based on randomization) begins on day 22 or when blood counts recover (whichever occurs later).

ARM B MAINTENANCE THERAPY: All patients receive vincristine sulfate IV over 1 minute on days 1, 29, and 57; dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61; mercaptopurine PO on days 1-84; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (omit day 29 for SR patients during the first 4 cycles); methotrexate IT on day 1 (and day 29 during the first 4 cycles for SR patients and during the first 2 cycles for IR patients). Patients with CNS1-3VHR and CNS2 VHR, and CNS3 IR disease also undergo cranial radiation therapy during the first 4 weeks (cycle 1). Treatment in female patients with T-ALL and patients with T-LLY repeats every 12 weeks for up to 2 years from the start of Interim Maintenance (week 119). Treatment in male patients with T-ALL repeats every 12 weeks for up to 3 years from the start of Interim Maintenance (week 171).

All treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* T-ALL: T-ALL patients must be enrolled on AALL08B1 or Project:EveryChild (APEC14B1, if open for the classification of ALL patients) prior to treatment and enrollment on AALL1231
* All patients must be > 1 and < 31 years of age
* Patients must have newly diagnosed T-lymphoblastic leukemia (T-ALL) or T-lymphoblastic lymphoma (T-LLy) stages II-IV

  * Note: a diagnosis of T-ALL is established when leukemic blasts lack myeloperoxidase or evidence of B-lineage derivation (cluster of differentiation [CD]19/CD22/CD20), and express either surface or cytoplasmic CD3 or two or more of the antigens CD8, CD7, CD5, CD4, CD2 or CD1a, and are present either in peripheral blood or > 25% in the bone marrow; if surface CD3 is expressed on all leukemic cells, additional markers of immaturity, including terminal deoxynucleotidyl transferase (TdT), CD34 or CD99 will be assessed for expression; cases with uncertain expression will receive additional review within the appropriate Children's Oncology Group (COG) reference laboratory
  * For T-LLy patients with tissue available for flow cytometry, the criterion for diagnosis should be analogous to T-ALL; for tissue processed by other means (i.e. paraffin blocks), the methodology and criteria for immunophenotypic analysis to establish the diagnosis of T-LLy defined by the submitting institution will be accepted
* All patients and/or their parents or legal guardians must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Patients must not have received any cytotoxic chemotherapy for either the current diagnosis of T-ALL, T-L-Ly or for any cancer diagnosis prior to the initiation of protocol therapy on AALL1231, with the exception of:

  * Steroid pretreatment: prednisone or methylprednisolone for =< 120 hours (5 days) in the 7 days prior to initiating induction chemotherapy or for =< 336 hours (14 days) in the 28 days prior to initiating induction chemotherapy; prior exposure to ANY steroids that occurred > 28 days before the initiation of protocol therapy does not affect eligibility; the dose of prednisone or methylprednisolone does not affect eligibility
  * Intrathecal cytarabine (the CNS status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment) system chemotherapy must begin with 72 hours of this IT therapy; or
  * Pretreatment with hydroxyurea; or
  * 600 cGy of chest irradiation, if medically necessary

    * Pre-treatment with dexamethasone in the 28 days prior to initiation of protocol therapy is not allowed with the exception of a single dose of dexamethasone use during sedation to prevent or treat airway edema; inhalation steroids and topical steroids are not considered pretreatment
* Pre-existing >= grade 2 sensory or motor peripheral neurotoxicity
* Uncontrolled seizure disorder
* Diagnosis of Down syndrome (Trisomy 21)
* Patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs; a pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* Patient has hypersensitivity to bortezomib, boron, or mannitol
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and within 30 days of any dose of bortezomib

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 847 (Actual)
Dates: Start 2014-10-04 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2026-09-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David T Teachey, Principal Investigator — Children's Oncology Group
Locations (212):
- United States (188):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Hayashi RJ, Hermiston ML, Wood BL, Teachey DT, Devidas M, Chen Z, Annett RD, Asselin BL, August K, Cho S, Dunsmore KP, Freedman JL, Galardy PJ, Harker-Murray P, Horton TM, Jaju A, Lam A, Messinger YH, Miles RR, Okada M, Patel S, Schafer ES, Schechter T, Shimano KA, Singh N, Steele A, Sulis ML, Vargas SL, Winter SS, Wood C, Zweidler-McKay PA, Loh ML, Hunger SP, Raetz EA, Bollard CM, Allen CE. MRD at the end of induction and EFS in T-cell lymphoblastic lymphoma: Children's Oncology Group trial AALL1231. Blood. 2024 May 16;143(20):2053-2058. doi: 10.1182/blood.2023021184. PMID 38457359
- [Derived] Gossai NP, Devidas M, Chen Z, Wood BL, Zweidler-McKay PA, Rabin KR, Loh ML, Raetz EA, Winick NJ, Burke MJ, Carroll AJ, Esiashvili N, Heerema NA, Carroll WL, Hunger SP, Dunsmore KP, Winter SS, Teachey DT. Central nervous system status is prognostic in T-cell acute lymphoblastic leukemia: a Children's Oncology Group report. Blood. 2023 Apr 13;141(15):1802-1811. doi: 10.1182/blood.2022018653. PMID 36603187
- [Derived] Teachey DT, Devidas M, Wood BL, Chen Z, Hayashi RJ, Hermiston ML, Annett RD, Archer JH, Asselin BL, August KJ, Cho SY, Dunsmore KP, Fisher BT, Freedman JL, Galardy PJ, Harker-Murray P, Horton TM, Jaju AI, Lam A, Messinger YH, Miles RR, Okada M, Patel SI, Schafer ES, Schechter T, Singh N, Steele AC, Sulis ML, Vargas SL, Winter SS, Wood C, Zweidler-McKay P, Bollard CM, Loh ML, Hunger SP, Raetz EA. Children's Oncology Group Trial AALL1231: A Phase III Clinical Trial Testing Bortezomib in Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia and Lymphoma. J Clin Oncol. 2022 Jul 1;40(19):2106-2118. doi: 10.1200/JCO.21.02678. Epub 2022 Mar 10. PMID 35271306
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Combination Chemotherapy): T-ALL; Arm A (Combination Chemotherapy): T-LLy: Patients receive combination chemotherapy without bortezomib.
- Arm B (Combination Chemotherapy, Bortezomib): T-ALL; Arm B (Combination Chemotherapy, Bortezomib): T-LLy: Patients received combination therapy with bortezomib (4 doses at 1.3mg/m2 during Induction and 4 doses at 1.3mg/m2 during Delayed Intensification)
Period: Overall Study
Arm/Group | Arm A (Combination Chemotherapy): T-ALL | Arm B (Combination Chemotherapy, Bortezomib): T-ALL | Arm A (Combination Chemotherapy): T-LLy | Arm B (Combination Chemotherapy, Bortezomib): T-LLy
Started | 312 | 315 | 111 | 109
Completed | 108 | 123 | 52 | 62
Not Completed | 204 | 192 | 59 | 47
Not completed — Adverse Event | 6 | 9 | 3 | 2
Not completed — Death | 9 | 9 | 3 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 94 | 72 | 24 | 15
Not completed — Withdrawal by Subject | 5 | 3 | 1 | 1
Not completed — Ineligible | 4 | 8 | 3 | 8
Not completed — Inevaluable | 6 | 4 | 5 | 5
Not completed — Refusal of further protocol therapy | 19 | 16 | 1 | 7
Not completed — Development of SMN | 1 | 0 | 0 | 1
Not completed — Relapse/Progression | 10 | 18 | 15 | 2
Not completed — VHR T-ALL who have an M2/M3 marrow and/or detectable MRD by end of the 3 HR Intensification Blocks | 5 | 5 | 0 | 0
Not completed — Still on Therapy | 44 | 47 | 3 | 2
Not completed — Identified to have Ph+ T-ALL | 0 | 1 | 0 | 0
Not completed — Identified to have Ph+ T-Lly | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Combination Chemotherapy): T-ALL | Arm B (Combination Chemotherapy, Bortezomib): T-ALL | Arm A (Combination Chemotherapy): T-LLy | Arm B (Combination Chemotherapy, Bortezomib): T-LLy | Total
Number analyzed (Participants) | 312 | 315 | 111 | 109 | 847
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 285 | 296 | 102 | 97 | 780
  Between 18 and 65 years | 27 | 19 | 9 | 12 | 67
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (5.7) | 10.1 (5.6) | 12.0 (5.3) | 12.3 (5.2) | 10.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 96 | 28 | 25 | 213
  Male | 248 | 219 | 83 | 84 | 634
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 62 | 17 | 15 | 146
  Not Hispanic or Latino | 236 | 228 | 86 | 89 | 639
  Unknown or Not Reported | 24 | 25 | 8 | 5 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 0 | 0 | 5
  Asian | 15 | 11 | 5 | 1 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 0 | 3
  Black or African American | 35 | 37 | 21 | 17 | 110
  White | 217 | 225 | 71 | 74 | 587
  More than one race | 6 | 6 | 1 | 0 | 13
  Unknown or Not Reported | 34 | 33 | 13 | 17 | 97
Region of Enrollment [Number; unit: participants]
  United States | 294 | 295 | 105 | 102 | 796
  Canada | 12 | 6 | 3 | 5 | 26
  Australia | 6 | 7 | 3 | 2 | 18
  New Zealand | 0 | 7 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) for Modified Augmented Berlin-Frankfurt-Munster Backbone With or Without Bortezomib in All Randomized Patients
Description: EFS is calculated as time from randomization at study entry to first event (induction failure, induction death, relapse, second malignancy, remission death) or date of last contact. Three-year EFS rates will be calculated for both groups.
Time Frame: 3 years
Population: As pre-specified in the protocol, this analysis includes all eligible patients (T-ALL+T-LLy) enrolled on the study. Arms were combined for this analysis as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Arm A (Combination Chemotherapy): Patients receive combination chemotherapy without bortezomib.
- Arm B (Combination Chemotherapy, Bortezomib): Patients received combination therapy with bortezomib (4 doses at 1.3mg/m2 during Induction and 4 doses at 1.3mg/m2 during Delayed Intensification)
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy, Bortezomib)
Number analyzed (Participants) | 416 | 408
Percentage of participants | 81.7 [77.0 to 86.4] | 85.1 [80.8 to 89.4]
Statistical Analysis 1: Comparison: Arm A (Combination Chemotherapy) vs Arm B (Combination Chemotherapy, Bortezomib); To compare the EFS of the randomized patients (T-ALL+T-LLy) on Arm A vs Arm B. Study was designed to accrue 1200 eligible, evaluable randomized patients (to provide 90.5% power to detect an improvement in 4-year EFS from 85% to 90% with an alpha of 0.05 (one-sided log-rank test) (Hazard Ratio (HR)=0.6483). Study was closed to accrual early due to results from AALL0434 for nelarabine; Test type: Superiority; p = 0.074, Log Rank; Hazard Ratio (HR) = 0.782, 95% CI 2-sided [0.561 to 1.091] — Hazard ratio = hazard rate for Arm B/hazard rate for Arm A

2. Secondary Outcome: Toxicity Rates Associated With Modified Standard Therapy, Including Dexamethasone and Additional Pegaspargase
Description: Percentage of patients who experienced Grade 3 or higher Toxicity Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: 3 years from start of therapy by patient
Population: As pre-specified in the protocol, this analysis includes all eligible patients (T-ALL+T-LLy) enrolled on the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Total Patients: All the eligible patients enrolled on the study
Arm/Group | Total Patients
Number analyzed (Participants) | 824
Percentage of participants | 78.0 [75.2 to 80.9]

3. Secondary Outcome: EFS for Standard (SR) and Intermediate Risk (IR) T-ALL Patients on the Non-bortezomib Containing Arm on This Study (no Cranial Radiation Therapy [CRT]) and Similar Patients on AALL0434 (Received CRT)
Description: EFS is calculated as time from randomization at study entry to first event (induction failure, induction death, relapse, second malignancy, remission death) or date of last contact.
Time Frame: 3 years
Population: T-ALL patients on AALL1231 who did not receive CRT or bortezomib: IR (exclude CNS3) and SR T-ALL (exclude those who met AALL0434 [NCT00408005] Low Risk definition). T-ALL on AALL0434 [NCT00408005] (who received CRT, no nelarabine) excluding Low Risk, CNS3, M3 Day 29, and EOC MRD >0.1%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- AALL1231 T-ALL Patients: T-ALL patients on AALL1231 who did not receive prophylactic cranial radiation and did not receive bortezomib: Intermediate Risk T-ALL (exclude CNS3) and SR T-ALL (exclude those who met AALL0434 Low Risk definition).
- AALL0434 T-ALL Patients: T-ALL patients on AALL0434 [NCT00408005] who received prophylactic cranial radiation and did not receive nelarabine (exclude Low Risk, CNS3, M3 Day 29, and EOC MRD >0.1%);
Arm/Group | AALL1231 T-ALL Patients | AALL0434 T-ALL Patients
Number analyzed (Participants) | 229 | 634
Percentage of participants | 88.3 [83.2 to 93.4] | 88.8 [86.3 to 91.4]

4. Secondary Outcome: Cumulative Incidence Rates of Isolated Central Nervous System (CNS) Relapse for SR and IR T-ALL Patients on the Non-bortezomib Containing Arm on This Study (no CRT) and Similar Patients on AALL0434 (Receive CRT)
Description: Cumulative incidence of isolated CNS relapse adjusting for competing risks using the method of: Gray R, A class of K-sample tests for comparing the cumulative incidence of a competing risk. Ann Stat 1141:1154, 1988
Time Frame: 3 years
Population: T-ALL patients on AALL1231 who did not receive CRT or bortezomib: IR (exclude CNS3) and SR T-ALL (exclude those who met AALL0434 [NCT00408005] Low Risk definition). T-ALL on AALL0434 [NCT00408005](who received CRT, no nelarabine) excluding Low Risk, CNS3, M3 Day 29, and EOC MRD >0.1%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AALL1231 T-ALL Patients | AALL0434 T-ALL Patients
Number analyzed (Participants) | 229 | 634
Percentage of participants
  Isolated CNS Relapse | 3.6 [1.1 to 6.1] | 2.2 [1.0 to 3.4]
  Isolated Bone Marrow Relapse | 1.4 [0 to 3.0] | 3.0 [1.6 to 4.4]
  Combined Bone Marrow Relapse | 1.3 [0 to 2.9] | 1.8 [0.8 to 2.8]

5. Secondary Outcome: EFS for Very High Risk (VHR) T-ALL Patients Treated With High Risk (HR) Berlin-Frankfurt-Munster (BFM) Intensification Blocks Who Become Minimal Residual Disease (MRD) Negative and Those Who Remain MRD Positive at the End of HR Block 3
Description: EFS will be calculated as time from the end of the three high-risk blocks of therapy to first event (relapse, second malignancy, remission death) or date of last contact.
Time Frame: 3 years
Population: VHR T-ALL patients who had EOC MRD >= 0.1%, completed the three high-risk blocks of therapy, and had MRD assessment done after the three high-risk blocks. MRD was not performed in T-LLy patients at end of the VHR blocks. MRD is not used in T-LLy to measure disease response. This outcome measure was pre-specified to only be assessed in the T-ALL patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- VHR T-ALL MRD Undetectable: VHR T-ALL patients (with end of consolidation [EOC] MRD >= 0.1%) who become MRD negative (MRD undetectable) after the three high-risk BFM blocks of therapy
- VHR T-ALL MRD Detectable: VHR T-ALL patients (with end of consolidation [EOC] MRD >= 0.1%) who continue to have detectable MRD after the three high-risk BFM blocks of therapy.
Arm/Group | VHR T-ALL MRD Undetectable | VHR T-ALL MRD Detectable
Number analyzed (Participants) | 8 | 10
Percentage of participants | 25.0 [0 to 67.5] | 88.9 [59.0 to 100]

6. Secondary Outcome: EFS for Very High Risk (VHR) T-LLy Patients Treated With HR Berlin-Frankfurt-Munster (BFM) Intensification Blocks Who Have Complete or Partial Remission and Those Who do Not Respond
Description: EFS for very high risk (VHR) T-LLy patients treated with HR Berlin-Frankfurt-Munster (BFM) intensification blocks who have complete or partial remission and those who do not respond
Time Frame: 3 years
Population: VHR T-LL patients who completed the three high-risk blocks of therapy. The T-LLy VHR patients are included in the table, but there were not enough patients to do any formal analysis, eg there was only one patient (n=1) on the study with T-LLy who had radiographic disease assessment after the intensification blocks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- VHR T-LLy (CR/PR): VHR T-LLy patients who achieved complete or partial response (CR/PR) at the end of the high-risk blocks
- VHR T-LLy (NR): VHR T-LLy patients who did not respond (NR) at the end of the high-risk blocks
Arm/Group | VHR T-LLy (CR/PR) | VHR T-LLy (NR)
Number analyzed (Participants) | 1 | 0
Percentage of participants | 0 |

ADVERSE EVENTS:
Time Frame: 3 years from start of therapy by patient
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm A (Combination Chemotherapy): T-ALL | Arm B (Combination Chemotherapy, Bortezomib): T-ALL | Arm A (Combination Chemotherapy): T-LLy | Arm B (Combination Chemotherapy, Bortezomib): T-LLy
All-Cause Mortality (participants affected / at risk) | 38/308 | 38/307 | 23/108 | 9/101
Serious Adverse Events (participants affected / at risk) | 56/308 | 153/307 | 25/108 | 60/101
Other Adverse Events (participants affected / at risk) | 231/308 | 217/307 | 86/108 | 74/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Combination Chemotherapy): T-ALL (N=308) | Arm B (Combination Chemotherapy, Bortezomib): T-ALL (N=307) | Arm A (Combination Chemotherapy): T-LLy (N=108) | Arm B (Combination Chemotherapy, Bortezomib): T-LLy (N=101)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (12) | 38 (51) | 2 (3) | 15 (20)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 10 (10) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 14 (16) | 5 (5) | 7 (9)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 6 (8) | 0 (0) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (2) | 3 (3)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 5 (5) | 0 (0) | 2 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 7 (7) | 1 (1) | 3 (3)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 5 (5) | 12 (15) | 1 (1) | 8 (10)
Lung infection (Infections and infestations) | 4 (4) | 5 (6) | 3 (3) | 3 (3)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 18 (20) | 26 (26) | 7 (7) | 11 (12)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (3)
Skin infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 14 (18) | 1 (1) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 6 (8) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 4 (4) | 15 (15) | 2 (2) | 2 (3)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 4 (4) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
INR increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 3 (3) | 7 (8) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
White blood cell decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 9 (10) | 1 (4) | 5 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 22 (25) | 2 (2) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 9 (10) | 1 (1) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 10 (11) | 1 (1) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (1) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 12 (12) | 1 (1) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Leukemia secondary to oncology chemotherapy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 5 (5)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 5 (5) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 1 (2) | 6 (7) | 0 (0) | 7 (7)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 6 (7) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (11) | 0 (0) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0) | 5 (5)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 2 (2) | 3 (3)
Pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 10 (11) | 1 (1) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2) | 17 (17) | 1 (1) | 6 (6)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Combination Chemotherapy): T-ALL (N=308) | Arm B (Combination Chemotherapy, Bortezomib): T-ALL (N=307) | Arm A (Combination Chemotherapy): T-LLy (N=108) | Arm B (Combination Chemotherapy, Bortezomib): T-LLy (N=101)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (20) | 25 (29) | 6 (11) | 7 (9)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (5) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 5 (5) | 1 (1) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 60 (68) | 56 (61) | 23 (25) | 24 (32)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 23 (30) | 29 (32) | 15 (20) | 11 (14)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 7 (7) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Death NOS (General disorders) | 16 (16) | 15 (15) | 10 (10) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 19 (19) | 12 (12) | 8 (8) | 1 (1)
Anaphylaxis (Immune system disorders) | 7 (8) | 10 (11) | 3 (3) | 6 (6)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 16 (17) | 24 (31) | 5 (6) | 5 (5)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 6 (6) | 3 (3) | 1 (1) | 4 (4)
Meningitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 31 (34) | 20 (20) | 10 (12) | 12 (14)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (5) | 1 (2) | 3 (3) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 11 (13) | 15 (21) | 5 (6) | 6 (11)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (5) | 2 (2) | 5 (5)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 42 (57) | 50 (78) | 20 (24) | 12 (17)
Cholesterol high (Investigations) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Fibrinogen decreased (Investigations) | 4 (5) | 3 (3) | 1 (1) | 1 (1)
GGT increased (Investigations) | 5 (5) | 7 (7) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 13 (16) | 13 (14) | 5 (6) | 4 (6)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6) | 10 (18) | 3 (5) | 2 (2)
Platelet count decreased (Investigations) | 3 (3) | 6 (8) | 1 (1) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 19 (22) | 18 (21) | 2 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6) | 6 (6) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 10 (15) | 13 (16) | 6 (7) | 7 (10)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (11) | 8 (8) | 4 (4) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 22 (25) | 21 (24) | 7 (9) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 50 (58) | 55 (59) | 21 (24) | 16 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 33 (39) | 26 (30) | 10 (13) | 12 (12)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 30 (47) | 25 (34) | 13 (17) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2) | 6 (7) | 3 (3)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 8 (8) | 2 (2) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 27 (30) | 26 (34) | 13 (16) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (32) | 27 (36) | 8 (10) | 7 (8)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 17 (19) | 10 (10) | 4 (8) | 6 (6)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 4 (4) | 4 (4) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 8 (8) | 6 (6) | 3 (3) | 3 (3)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 13 (14) | 7 (7) | 11 (13) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT02112916/Prot_SAP_000.pdf